CLINICAL TRIAL: NCT02945761
Title: Ningbo NO.4 Hospital,CHINA.
Brief Title: High Concentration of Sugar Solution Irrigation Promotes the Healing of Infected Wound
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Ningbo Municipal No.4 Hospital (Other Government)
Responsible Party: Principal Investigator, weng xinhai, Director, Ningbo Municipal No.4 Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: wengxinhai
Record Dates: First submitted 2016-10-23; First posted 2016-10-26 (Estimated); Last update posted 2016-10-26 (Estimated); Status verified 2016-10

CONDITIONS: Wound Infection; Sugar Solution
MeSH Terms: conditions — Wound Infection

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (2):
- High concentration of sugar solution (Active Comparator): Lavage group of high-concentration sugar solution (HCSS): disinfected the Skin outside wound with conventional PVP. HCSS refers to supersaturated sugar solution made of 50% high-concentration glucose and white sugar. Prior to wound irrigation, dry cotton balls are used to wipe the wound and internal lacuna, to clean some necrotic tissues out of the wound. HCSS is applied on the wound once a day, and whether the lavaging is stopped based on the amount of exudation from the wound.
  Interventions: Procedure: High concentration of sugar solution
- conventional surgical dressing change (Active Comparator): conventional surgical dressing change:separated suture, expanded the wound, placed drainage ribbon gauze and used hydrogen peroxide or(and) PVP to wash the wound; the decision-making power of these operators is determined by a doctor. After the doctor confirms granulation cleaning in the wound, the decision-making power of suture is also determined by a doctor.
  Interventions: Procedure: conventional surgical dressing change

INTERVENTIONS:
Procedure: High concentration of sugar solution
  Arms: High concentration of sugar solution
Procedure: conventional surgical dressing change
  Arms: conventional surgical dressing change

SUMMARY:
Surgeons easily get wound infections. Most wound infections will be cured by applying medicines and changing dressing in very short period of time. But some wounds are severely contaminated combined with fat liquefaction, crateriform ulcer and large undermined lacuna, so changing dressing takes a very long time. In order to better change the dressing, it needs to expose the wound thoroughly, which requires to completely open the healed skin, so the healing will be slowed down. Some scholars lay stress on prevention. Wound infection control concerns prevention--not therapy--of an infrequent but expensive kind of surgical morbidity.(1.2)Some scholars think that the main armamentarium of the attack is the use of topical anti-infectives, which invade the bacteria where they reside, and, consequently, reduce their numbers and promote wound healing.(3)For example, silver is reemerging as a viable treatment option for infections encountered in burns, open wounds, and chronic ulcers. But it is expensive and is difficult to acquire silver-containing dressings. And Recent findings, however, indicate that the compound delays the wound-healing process and that silver may have serious cytotoxic activity on various host cells. (4) As High concentration of sugar solution, honey appears to heal partial thickness burns more quickly than conventional treatment (which included polyurethane film, paraffin gauze, soframycin-impregnated gauze, sterile linen and leaving the burns exposed) and infected post-operative wounds more quickly than antiseptics and gauze.(5)This study involve the use of another high-concentration of sugar solution (HCSS) to lavage infected wounds when changing dressings.

ELIGIBILITY:
Inclusion Criteria:

1. Patients conducted surgical operation in the hospital within 2 weeks. The wound had swelling and lots of secretions;
2. Except for the incision, primary surgical site has been recovered smoothly. Patients didn't accept secondary operation in the same site;

Exclusion Criteria:

1. Except for the wound that can't use healthy skin closure in Phase I

Ages: 1 Year to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 3 (Estimated)
Dates: Start 2016-10; Primary Completion 2017-10 (Estimated)

PRIMARY OUTCOMES:
Duration of wound healing | 4 weeks
  It means the time from the first day after incision infection is found out to continuous dressing change in the last time. If the wound is kept in the infection status, it requires changing it for the wound once a day. For phase II suture on the open incision, the last time of dressing change should add the following days. Abdominal incision should increase 5 days. The wound of four limbs should increase 10 days.
The scoring on the open wound | 4 weeks
  Without separating suture, only the wound is shoved off within 2cm for 1 score; with separating suture, but the distance is kept in 2cm for 2 scores; with separating suture, the wound is shoved off for 2-3cm for 3 scores; In a similar fashion, the highest one is 10 scores. For patients with the longer wound and disconnected openness, the overall length of the wound should be overlapped. According to the overall length, scores are conducted as the above-mentioned rules.

CONTACTS AND LOCATIONS:
Overall Officials: xinhai weng, BS, Study Director — Ningbo NO.4 hospital